CLINICAL TRIAL: NCT00768547
Title: Risk Stratification in Acutely Admitted Medical Patients
Status: Completed | Type: Observational
Sponsor: Ribe County Hospital (Other)
Responsible Party: MIkkel Brabrand, MD, Ribe County Hospital
Other Study IDs: risk stratification
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2008-08

CONDITIONS: Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- By protocol: Where the test are predefined
- By degression: The group where the doctor decided which test are to be taken.

SUMMARY:
The study has three main parts.

1. To see if we can develop a riskstratification tool that can be used to asses the risk for acutely admitted medical patients for inhospital death, admission to the ICU and death within 30 days of release.
2. To test existing tool as in 1.
3. To clarify if it is most reasonable to let the admitting doctor order blood test by clinical judgment or be using a predefined list of tests.

ELIGIBILITY:
Inclusion Criteria:

* Any patient acutely admitted to the medical department of Ribe County Hospital

Exclusion Criteria:

* Age below 15 years
* Unwilling to participate

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient acutely admitted to the medical department of Ribe County Hospital
Sampling Method: Non-Probability Sample
Enrollment: 5900 (Actual)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of test taken in each group | Five months

CONTACTS AND LOCATIONS:
Locations (1):
- Ribe County Hospital, Esbjerg, Esbjerg, Denmark